CLINICAL TRIAL: NCT01875757
Title: Effect of Supplementation With Vitamin D on the Acute Bronchitis Prevention During the First Year of Life
Acronym: VitDBR2012
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012-001152-19; 2012-001152-19 (EudraCT Number)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Acute Bronchitis; Upper Respiratory Tract Infection; Acute Bronchiolitis
Keywords: Vitamin D; Acute bronchitis; Upper respiratory tract infection; Recurrent bronchitis; Acute bronchiolitis; Infants
MeSH Terms: conditions — Bronchitis; Respiratory Tract Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Vitamin D3 1000 IU/day (Experimental): Infants will be supplemented with vitamin D and/or placebo to receive a total amount of vitamin D3 of 1.000 IU/day during the first year of life, taking into account the vitamin D received with artificial milk
  Interventions: Drug: Vitamin D3; Drug: Placebo
- Vitamin D3 400 IU/day (Active Comparator): Infants will be supplemented with vitamin D and/or placebo to receive a total amount of vitamin D3 of 400 IU/day during the first year of life, taking into account the vitamin D received with artificial milk
  Interventions: Drug: Vitamin D3; Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3
Drug: Placebo

SUMMARY:
A phase III multicenter randomized double blind clinical trial will be conducted. After obtaining written consent the infant will be randomized, during the first two weeks of life, to a study group to receive either 400 IU or 1,000 IU / day of vitamin D to the year of age.

Baseline and all follow up visits (2, 6, and 12 months of life) will include anthropometric measurements and a questionnaire about health issues. A blood sample will be obtained at baseline for analysis of 25OH vitamin D, and at 6 and 12 months for analysis of 25 OH vitamin D, and calcium.

Healthy term born infants of appropriate size for gestational age will be included. We will need to include 359 children in each group.

The primary objective of the study is to decrease the proportion of infants with acute bronchitis during the first year of life by supplementation of 1,000 IU/day vitamin D. Secondary otcomes are: To check that the administration of 1,000 IU/day vitamin D decreases the proportion of infants with upper respiratory tract infections, the proportion of children under one year of age hospitalized for acute bronchiolitis, and the demand on the healthcare system due to respiratory infections and absences from work for parents and achieves a higher proportion of children with adequate blood levels 25 OH vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term born infants of appropriate size for gestational age
* Parents provide informed consent to participate

Exclusion Criteria:

* Infants with small size for gestational age
* Infants with gestational age < 37 weeks
* Infants with congenital anomalies
* Infants with chronic gastrointestinal tract, liver, kidney, heart, or neurological diseases
* Infants with disorders of vitamin D or calcium metabolism or others inborn errors of metabolism

Max Age: 19 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of children with acute bronchitis | 1 year
  Check that the administration of a vitamin D dose of 1,000 U / day decreases the percentage of children with acute bronchitis during the first year of life

SECONDARY OUTCOMES:
Number of episodes of upper respiratory infections reported by parents in the first year of life | 1 year
  Check that the supplementation of vitamin D of 1,000 units / day decreases the number of upper respiratory infections

OTHER OUTCOMES:
Percentage of children with recurrent bronchitis | 1 year
  Check that the supplementation of vitamin D of 1,000 units / day decreases the number of recurrent bronchitis

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Moreno, MD, PhD, Study Chair — Hospital Universitari Vall d'hebron Barcelona, Spain
Locations (1):
- Hospital Universitary Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Camargo CA Jr, Ingham T, Wickens K, Thadhani R, Silvers KM, Epton MJ, Town GI, Pattemore PK, Espinola JA, Crane J; New Zealand Asthma and Allergy Cohort Study Group. Cord-blood 25-hydroxyvitamin D levels and risk of respiratory infection, wheezing, and asthma. Pediatrics. 2011 Jan;127(1):e180-7. doi: 10.1542/peds.2010-0442. Epub 2010 Dec 27. PMID 21187313
- [Background] Belderbos ME, Houben ML, Wilbrink B, Lentjes E, Bloemen EM, Kimpen JL, Rovers M, Bont L. Cord blood vitamin D deficiency is associated with respiratory syncytial virus bronchiolitis. Pediatrics. 2011 Jun;127(6):e1513-20. doi: 10.1542/peds.2010-3054. Epub 2011 May 9. PMID 21555499
- [Background] Karatekin G, Kaya A, Salihoglu O, Balci H, Nuhoglu A. Association of subclinical vitamin D deficiency in newborns with acute lower respiratory infection and their mothers. Eur J Clin Nutr. 2009 Apr;63(4):473-7. doi: 10.1038/sj.ejcn.1602960. Epub 2007 Nov 21. PMID 18030309
- [Background] Urashima M, Segawa T, Okazaki M, Kurihara M, Wada Y, Ida H. Randomized trial of vitamin D supplementation to prevent seasonal influenza A in schoolchildren. Am J Clin Nutr. 2010 May;91(5):1255-60. doi: 10.3945/ajcn.2009.29094. Epub 2010 Mar 10. PMID 20219962
- [Background] Devereux G, Litonjua AA, Turner SW, Craig LC, McNeill G, Martindale S, Helms PJ, Seaton A, Weiss ST. Maternal vitamin D intake during pregnancy and early childhood wheezing. Am J Clin Nutr. 2007 Mar;85(3):853-9. doi: 10.1093/ajcn/85.3.853. PMID 17344509
- [Background] Camargo CA Jr, Rifas-Shiman SL, Litonjua AA, Rich-Edwards JW, Weiss ST, Gold DR, Kleinman K, Gillman MW. Maternal intake of vitamin D during pregnancy and risk of recurrent wheeze in children at 3 y of age. Am J Clin Nutr. 2007 Mar;85(3):788-95. doi: 10.1093/ajcn/85.3.788. PMID 17344501